CLINICAL TRIAL: NCT01464684
Title: Body Composition of Infants: Follow-up to Placenta and Cord Blood Analyses
Status: Withdrawn | Type: Observational
Why Stopped: determined not enough participants would be able to be enrolled and not enough data collected for good analyses
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 132624
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Infant Body Composition and Metabolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, and a cheek swab may be collected from study participants

SUMMARY:
Investigators will characterize the body composition and metabolism of infants born from lean, overweight or obese mothers from whom they had previously obtained a placenta and/or cord blood as part of the earlier placenta and cord blood study (#111576)

ELIGIBILITY:
Inclusion Criteria:

* mother's prior participation in study #111576 with successful collection of placenta
* infant age 12 months (+/- 9 months)

Exclusion Criteria:

* mother did not participate in study #111576
* mother did participate in study #111576, but collection of placenta was not successful
* infant not age 12 months (+/- 9 months)

Ages: 3 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infants age 12 months (+/- 9 months)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Aline Andres, PhD, Principal Investigator — University of Arkansas